CLINICAL TRIAL: NCT03515785
Title: A Postmarketing Observational Cohort Study to Evaluate Effectiveness and Safety of Ponatinib (Iclusig®) in Patients With BCR-ABL Positive ALL in Standard Clinical Practice in Europe - "POSEIDON"
Brief Title: A Study to Evaluate Effectiveness and Safety of Ponatinib in Patients With BCR-ABL Positive ALL in Standard Clinical Practice in Europe - "POSEIDON"
Status: Withdrawn | Type: Observational
Why Stopped: Revisiting the availability of patients with Ph+ ALL that would meet the in-/exclusion criteria of the study led to the decision not to move forward.
Sponsor: Incyte Biosciences International Sàrl (Industry)
Responsible Party: Sponsor
Organization: Incyte Corporation (Industry)
Other Study IDs: INCB-DEMA-ALL-401
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: BCR-ABL Positive Acute Lymphoblastic Leukemia
Keywords: acute lymphoblastic leukemia; ponatinib; tyrosine kinase inhibitor
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ph+ ALL Patients: Patients with Ph+ ALL being treated with Iclusig®.

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of ponatinib (Iclusig®) in patients with BCR-ABL positive acute lymphoblastic leukemia (ALL) in standard clinical practice in Europe.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with BCR-ABL (Ph+) positive ALL who are initiating Iclusig®, or for whom Iclusig® was initiated after January 2015.
* Patients who have the ability to understand the requirements of the study and provide written informed consent to comply with the study data collection procedures.

Exclusion Criteria:

* Patients previously treated with investigational ponatinib.
* Patients who are pregnant and/or breastfeeding.
* Concurrent treatment with another tyrosine kinase inhibitor for Ph+ALL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Ph+ ALL being treated with Iclusig® in Europe.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-12-31 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Complete hematological remission (CR) rate | 6 months
  CR defined as leukemic cells not detectable by light microscopy in bone marrow (BM), peripheral blood (PB), or cerebrospinal fluid (CSF) (BM < 5% blasts).

SECONDARY OUTCOMES:
CR rate | 1, 3, 9, and 12 months
  CR defined as leukemic cells not detectable by light microscopy in BM, PB, or CSF (BM < 5% blasts).
CR rate | 1, 3, 6, 9, and 12 months
  CR defined as leukemic cells not detectable by light microscopy in BM, PB, or CSF (BM < 5% blasts).
Time to CR | Up to 12 months
  Defined as time from enrollment to first CR.
Minimal residual disease (MRD) level | 3, 6, 9, and 12 months
  Minimal residual disease level.
Best MRD (MolR) level rate | 12 months
  MolR defined as molecular/MRD response, less than MolCR.
Time to best MRD (MolR) level | Up to 12 months
  MolR defined as molecular/MRD response, less than MolCR.
Duration of molecular response | Up to 12 months
  Measured by MRD log reduction (MolR).
Duration of best molecular response (MolCR) | Up to 12 months
  MolCR defined as complete molecular remission/MRD negativity.
Time to progression | Up to 12 months
  Defined as the time to molecular relapse or hematological relapse.
Time to death | Up to 12 months
  Defined as time from enrollment to death due to any cause.
Prescribed dose | Up to 12 months
  Prescribed dose of Iclusig® in milligrams.
Daily average dose | Up to 12 months
  The average daily dose of Iclusig® in milligrams.
Number of serious adverse events (SAEs) | 12 months
  Defined as an adverse event that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Number of adverse events of special interest (AESI) | 12 months
  AESI defined as vascular occlusive events, including arterial and venous events, as defined in the protocol.
Amount of hospital days | 12 months
  Defined as overnight stay(s), each night in the hospital will be counted as 1 day.

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Hoelzer, Prof. Dr. med., Principal Investigator — Oncologikum Frankfurt
Locations (10):
- Ihbt/Úhkt, Prague, Czechia
- France (6):
  - University Hospital Amiens, Amiens
  - University Hospital Angers, Angers
  - University Hospital Bordeaux, Bordeaux
  - University Hospital Grenoble, Grenoble
  - University Hospital Lyon, Lyon
  - University Cancer Institute Oncopole, Toulouse
- Germany (3):
  - University Hospital Halle/Saale, Halle
  - University Hospital Munich, Munich
  - University Hospital Rostock, Rostock

IPD SHARING:
Plan to Share IPD: No